CLINICAL TRIAL: NCT01760187
Title: A Randomized, Double-blind, Placebo-controlled, Single Ascending and Multiple Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics(PK) and Pharmacodynamics(PD) of Lomitapide in Japanese and Caucasian Volunteers With Elevated Low-density-lipoprotein(LDL-C)
Brief Title: Phase I Study of the Safety, Tolerability, PK & PD of Lomitapide in Japanese and Caucasian Subjects With Elevated LDL-C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aegerion Pharmaceuticals, Inc. (Industry)
Collaborators: Richmond Pharmacology Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AEGR-733-023; 2012-004220-37 (EudraCT Number)
Record Dates: First submitted 2012-11-21; First posted 2013-01-04 (Estimated); Results first posted 2018-11-20 (Actual); Last update posted 2018-11-20 (Actual); Status verified 2018-11

CONDITIONS: Healthy Volunteer
MeSH Terms: interventions — BMS201038

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Cohort 1 (Experimental): 12 Japanese and 12 Caucasian subjects. 10 out of 12 will receive 10 mg lomitapide and 2 will receive placebo.
  Interventions: Drug: lomitapide
- Cohort 2 (Experimental): 8 Japanese and 8 Caucasian subjects. 6 out of 8 subjects will receive 20 mg lomitapide and 2 will receive placebo.
  Interventions: Drug: lomitapide
- Cohort 3 (Experimental): 8 Japanese and 8 Caucasian subjects. 6 out of 8 subjects will receive 40 mg lomitapide and 2 will receive placebo.
  Interventions: Drug: lomitapide
- Cohort 4 (Experimental): 8 Japanese and 8 Caucasian subjects. 6 out of 8 subjects will receive 60 mg lomitapide and 2 will receive placebo.
  Interventions: Drug: lomitapide

INTERVENTIONS:
Drug: lomitapide

SUMMARY:
This is a randomized, double-blind, placebo-controlled, single ascending dose (SAD) and multiple ascending dose (MAD) study of orally administered lomitapide in healthy male Japanese and Caucasian subjects with elevated LDL-C. The purpose for this study is to evaluate the PK and PD of lomitapide in Japanese subjects as compared to Caucasian subjects.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject is a healthy male or female, Caucasian or Japanese, aged 20 - 45 years, inclusive, at screening.

  2. Subject has a BMI of 18.5 - 30 kg/m2 inclusive at screening.

  3. Subjects must have a screening LDL-C measurement and the mean of Day 5 and Day 6 measurements greater than or equal to 110mg/dL.

  4. Subjects must agree to use acceptable methods of contraception (details provided in the protocol)

  5. Subjects must be capable of understanding and complying with the requirements of the protocol and must have signed the informed consent form prior to undergoing any study-related procedures.

Exclusion Criteria:

1. Subject has a clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion.
2. Any clinically significant abnormal laboratory, vital signs or other safety findings as determined by medical history, physical examination or other evaluations conducted at screening or on admission.
3. Electrocardiogram (ECG) abnormalities in the standard 12-lead ECG (at screening) which in the opinion of the Investigator is clinically relevant or will interfere with the ECG analysis.
4. History or current evidence of any clinically relevant cardiovascular, pulmonary, hepatic, renal, gastrointestinal, haematological, endocrinological, metabolic, neurological, psychiatric or other disease.
5. Positive results in any of the serology tests for Hepatitis B Surface Antigen (HbsAg), anti-Hepatitis core antibody (anti-HBc Ig G [and anti-HBc IgM if IgG is positive], Hepatitis C antibodies (anti-HCV), and HIV 1 and 2 antibodies, (anti-HIV 1/2) at screening.
6. Confirmed positive results from urine drug screen or from the alcohol breath test at screening and on admission (Day -1).
7. History or clinical evidence of alcohol or drug abuse.
8. Mentally handicapped.
9. Participation in a drug trial within 90 days prior to first drug administration.
10. Use of any medication (including over-the-counter (OTC) medication) within 2 weeks prior to admission (Day -1) or within less than 10 times the elimination half-life of the respective drug, or anticipated concomitant medication during the treatment periods.
11. Use of any substance inhibiting CYP3A4 enzymes within 2 weeks prior to admission (Day -1).
12. Donation of more than 500 mL of blood within 90 days prior to drug administration.
13. Subjects who smoke more than 10 cigarettes or equivalent amount of tobacco per day and/or who cannot stop smoking for the duration of the study whilst in the CPU.
14. Treatment with herbal supplements during the 7 days prior to dosing, or use of vitamins during 48 hours prior to admission (Day -1).
15. Any circumstances or conditions, which, in the opinion of the PI, may affect full participation in the trial or compliance with the protocol.
16. Legal incapacity or limited legal capacity at screening.
17. Subjects who are vegetarians, vegans or have any dietary restrictions conflicting with the study standardised menus.
18. If female, subject was pregnant or lactating (females of child bearing potential must have negative pregnancy tests at screening and admission).

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2012-11-07 (Actual); Primary Completion 2013-06-03 (Actual); Study Completion 2013-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Lorch, MD FRCA FFPM, Principal Investigator — Richmond Pharmacology Limited
Locations (1):
- Richmond Pharmacology Ltd, Croydon, Surrey, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: 10 Japanese and 10 Caucasian subjects will receive 10 mg lomitapide.
- Cohort 2: 6 Japanese and 6 Caucasian subjects will receive 20 mg lomitapide.
- Cohort 3: 6 Japanese and 6 Caucasian subjects will receive 40 mg lomitapide.
- Cohort 4: 6 Japanese and 6 Caucasian subjects will receive 60 mg lomitapide.
- Placebo: 8 Japanese and 8 Caucasian subjects will receive placebo.
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Placebo
Started | 20 | 12 | 12 | 12 | 16
Completed | 19 | 12 | 12 | 10 | 16
Not Completed | 1 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo - Japanese Patients: 8 Japanese patients will receive placebo, across the cohorts.
  (2 at each cohort)
- Placebo - Caucasian Patients: 8 Caucasian patients will receive placebo, across the cohorts.
  (2 at each cohort)
- Cohort 1- Japanese Patients: 10 Japanese subjects will receive 10 mg of lomitapide.
- Cohort 1 - Caucasian Patients: 10 Caucasian subjects will receive 10 mg of lomitapide.
- Cohort 2 - Japanese Patients: 6 Japanese subjects will receive 20 mg of lomitapide.
- Cohort 2 - Caucasian Patients: 6 Caucasian subjects will receive 20 mg of lomitapide.
- Cohort 3 - Japanese Patients: 6 Japanese subjects will receive 40 mg of lomitapide.
- Cohort 3 - Caucasian Patients: 6 Caucasian subjects will receive 40 mg of lomitapide.
- Cohort 4 - Japanese Patients: 6 Japanese subjects will receive 60 mg of lomitapide.
- Cohort 4 - Caucasian Patients: 6 Caucasian subjects will receive 60 mg of lomitapide.
- Total: Total of all reporting groups
Arm/Group | Placebo - Japanese Patients | Placebo - Caucasian Patients | Cohort 1- Japanese Patients | Cohort 1 - Caucasian Patients | Cohort 2 - Japanese Patients | Cohort 2 - Caucasian Patients | Cohort 3 - Japanese Patients | Cohort 3 - Caucasian Patients | Cohort 4 - Japanese Patients | Cohort 4 - Caucasian Patients | Total
Number analyzed (Participants) | 8 | 8 | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 72
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.1 (6.0) | 33.6 (7.3) | 33.8 (6.0) | 31.2 (6.6) | 32.2 (5.4) | 36.0 (7.5) | 32.5 (4.6) | 31.2 (9.7) | 30.2 (5.4) | 37.7 (3.4) | 33.3 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 8 | 8 | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 72
Region of Enrollment [Number; unit: participants]
  United Kingdom | 8 | 8 | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6 | 72

OUTCOME MEASURES:

1. Primary Outcome: Cmax for Lomitapide
Description: Maximum observed plasma concentration for lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 7
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Japanese 10 mg: Japanese Subjects who received 10 mg Lomitapide
- Caucasian 10 mg: Caucasian Subjects who received 10 mg Lomitapide
- Japanese 20 mg: Japanese Subjects who received 20 mg Lomitapide
- Caucasian 20 mg: Caucasian Subjects who received 20 mg Lomitapide
- Japanese 40 mg: Japanese Subjects who received 40 mg Lomitapide
- Caucasian 40 mg: Caucasian Subjects who received 40 mg Lomitapide
- Japanese 60 mg: Japanese Subjects who received 60 mg Lomitapide
- Caucasian 60 mg: Caucasian Subjects who received 60 mg Lomitapide
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 0.570 (0.285) | 0.436 (0.166) | 1.70 (0.49) | 1.01 (0.17) | 3.93 (0.75) | 3.00 (1.52) | 8.29 (3.44) | 5.75 (1.78)

2. Primary Outcome: Tmax for Lomitapide
Description: Time to maximum observed concentration for lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 7
Population: All subjects with evaluable concentrations
Measure: Median (Full Range); unit: hr
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
hr | 4 [2 to 6] | 5 [2 to 12] | 9 [4 to 12] | 6 [2 to 12] | 4 [2 to 6] | 5 [4 to 8] | 6 [4 to 6] | 5 [2 to 6]

3. Primary Outcome: AUC0-t for Lomitapide
Description: Area under the plasma concentration versus time curve from hour 0 to the last measurable concentration for lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 7
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 29.1 (13.0) | 27.5 (11.0) | 63.0 (16.0) | 54.2 (9.6) | 152 (48) | 123 (53) | 238 (84) | 241 (72)

4. Primary Outcome: AUC0-∞ for Lomitapide
Description: Area under the plasma concentration versus time curve from zero to infinity for lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 7
Population: AUC0-∞ and t1/2 were not calculated for 3 subjects in the Japanese 10mg arm because the estimated t1/2 was being much longer than half of the total sampling time.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 7 | 10 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 37.3 (16.7) | 35.9 (15.3) | 68.6 (17.4) | 64.7 (14.7) | 168 (59) | 133 (58) | 251 (89) | 260 (74)

5. Primary Outcome: t1/2 for Lomitapide
Description: Apparent terminal elimination half-life for lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 7
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 7 | 10 | 6 | 6 | 6 | 6 | 6 | 6
hr | 79.5 (5.6) | 82.8 (5.9) | 50.5 (2.6) | 64.3 (20.6) | 58.8 (13.3) | 56.2 (7.1) | 44.9 (5.7) | 51.5 (10.9)

6. Primary Outcome: Cmax for Lomitapide
Description: Maximum observed plasma concentration for lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 27
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 2.46 (0.88) | 3.31 (2.91) | 5.96 (2.79) | 4.35 (1.07) | 19.7 (6.2) | 13.8 (5.1) | 29.6 (11.1) | 24.6 (9.0)

7. Primary Outcome: Tmax for Lomitapide
Description: Time to maximum observed concentration for lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 27
Population: All subjects with evaluable concentrations
Measure: Median (Full Range); unit: hr
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
hr | 4 [1 to 4] | 4 [2 to 6] | 4 [1 to 8] | 4 [4 to 4] | 4 [4 to 4] | 4 [4 to 6] | 4 [2 to 6] | 4 [2 to 4]

8. Primary Outcome: AUC0-t for Lomitapide
Description: Area under the plasma concentration versus time curve from hour 0 to the last measurable concentration for lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 27
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 38.1 (14.1) | 44.5 (29.0) | 91.3 (29.5) | 74.4 (18.8) | 263 (64) | 204 (79) | 388 (86) | 403 (130)

9. Primary Outcome: t1/2 for Lomitapide
Description: Apparent terminal elimination half-life for lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 27
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
hr | 62.6 (10.1) | 57.6 (8.9) | 56.1 (9.9) | 53.3 (8.5) | 49.7 (11.3) | 44.8 (6.4) | 48.9 (9.9) | 46.5 (6.3)

10. Secondary Outcome: Cmax for M1
Description: Maximum observed plasma concentration for M1 metabolite of lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 7
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 1.23 (0.23) | 1.02 (0.23) | 2.27 (0.54) | 1.86 (0.54) | 4.18 (1.22) | 4.20 (1.72) | 7.43 (1.88) | 5.53 (0.83)

11. Secondary Outcome: Tmax for M1
Description: Time to maximum observed concentration for M1 metabolite of lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 7
Population: All subjects with evaluable concentrations
Measure: Median (Full Range); unit: hr
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
hr | 6 [4 to 8] | 6 [4 to 6] | 5 [4 to 6] | 6 [4 to 8] | 4 [1 to 8] | 6 [4 to 8] | 6 [4 to 6] | 6 [2 to 8]

12. Secondary Outcome: AUC0-t for M1
Description: Area under the plasma concentration versus time curve from hour 0 to the last measurable concentration for M1 metabolite of lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 7
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 37.1 (9.7) | 32.1 (7.9) | 64.1 (15.6) | 56.7 (18.6) | 134 (37) | 129 (57) | 199 (64) | 177 (44)

13. Secondary Outcome: AUC0-∞ for M1
Description: Area under the plasma concentration versus time curve from zero to infinity for M1 metabolite of lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 7
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 38.7 (10.1) | 34.0 (8.3) | 65.7 (15.9) | 59.1 (19.5) | 138 (39) | 132 (58) | 204 (67) | 183 (46)

14. Secondary Outcome: t1/2 for M1
Description: Apparent terminal elimination half-life for M1 metabolite of lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 7
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
hr | 37.8 (11.3) | 44.0 (14.3) | 35.9 (8.7) | 35.9 (6.0) | 41.5 (4.3) | 36.3 (7.9) | 39.4 (3.4) | 43.6 (4.9)

15. Secondary Outcome: Cmax for M3
Description: Maximum observed plasma concentration for M3 metabolite of lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 7
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 20.0 (4.1) | 14.2 (4.8) | 35.3 (8.2) | 20.0 (5.8) | 55.7 (18.3) | 50.9 (24.7) | 83.9 (34.5) | 67.7 (23.8)

16. Secondary Outcome: Tmax for M3
Description: Time to maximum observed concentration for M3 metabolite of lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 7
Population: All subjects with evaluable concentrations
Measure: Median (Full Range); unit: hr
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
hr | 4 [2 to 4] | 3 [2 to 4] | 4 [2 to 4] | 4 [2 to 4] | 3 [1 to 4] | 2 [2 to 4] | 4 [4 to 4] | 2 [1 to 4]

17. Secondary Outcome: AUC0-t for M3
Description: Area under the plasma concentration versus time curve from hour 0 to the last measurable concentration for M3 metabolite of lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 7
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 265 (53) | 185 (86) | 486 (145) | 263 (115) | 760 (169) | 824 (355) | 1410 (675) | 1170 (541)

18. Secondary Outcome: AUC0-∞ for M3
Description: Area under the plasma concentration versus time curve from zero to infinity for M3 metabolite of lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 7
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 276 (55) | 196 (91.2) | 501 (147) | 274 (119) | 780 (171) | 839 (361) | 1430 (693) | 1200 (551)

19. Secondary Outcome: t1/2 for M3
Description: Apparent terminal elimination half-life for M3 metabolite of lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 7
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
hr | 56.3 (11.6) | 56.9 (10.2) | 53.1 (12.9) | 51.3 (6.4) | 50.5 (14.9) | 39.4 (6.1) | 47.0 (7.4) | 43.8 (5.3)

20. Secondary Outcome: Cmax for M1
Description: Maximum observed plasma concentration for M1 metabolite of lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 27
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 2.56 (0.44) | 2.15 (0.53) | 4.36 (0.88) | 4.24 (1.30) | 9.98 (4.13) | 10.7 (3.6) | 13.5 (3.4) | 12.6 (3.2)

21. Secondary Outcome: Tmax for M1
Description: Time to maximum observed concentration for M1 metabolite of lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 27
Population: All subjects with evaluable concentrations
Measure: Median (Full Range); unit: hr
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
hr | 6 [2 to 8] | 6 [2 to 6] | 6 [4 to 6] | 6 [4 to 8] | 4 [4 to 8] | 6 [4 to 6] | 6 [4 to 8] | 4 [4 to 8]

22. Secondary Outcome: AUC0-t for M1
Description: as for outcome 12
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 27
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 44.3 (8.5) | 36.1 (8.5) | 73.7 (14.4) | 75.3 (25.9) | 180 (78) | 176 (58) | 230 (71) | 223 (66)

23. Secondary Outcome: t1/2 for M1
Description: Apparent terminal elimination half-life for M1 metabolite of lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 27
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
hr | 42.4 (9.0) | 41.9 (7.5) | 41.6 (8.5) | 39.7 (4.5) | 41.0 (6.6) | 36.0 (1.7) | 43.5 (7.8) | 41.2 (6.2)

24. Secondary Outcome: Cmax for M3
Description: Maximum observed plasma concentration for M3 metabolite of lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 27
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
ng/mL | 33.9 (9.3) | 24.1 (7.9) | 56.4 (15.0) | 35.2 (18.8) | 76.3 (26.7) | 86.4 (27.1) | 129 (35) | 126 (50)

25. Secondary Outcome: Tmax for M3
Description: Time to maximum observed concentration for M3 metabolite of lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 27
Population: All subjects with evaluable concentrations
Measure: Median (Full Range); unit: hr
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
hr | 2 [2 to 4] | 3 [2 to 6] | 3 [2 to 4] | 4 [2 to 4] | 4 [2 to 4] | 4 [2 to 6] | 4 [2 to 6] | 2 [2 to 4]

26. Secondary Outcome: AUC0-t for M3
Description: as for outcome 17
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 27
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
ng*hr/mL | 335 (84) | 239 (90) | 617 (163) | 386 (183) | 891 (259) | 1150 (462) | 1640 (664) | 1640 (767)

27. Secondary Outcome: t1/2 for M3
Description: Apparent terminal elimination half-life for M3 metabolite of lomitapide
Time Frame: 1, 2, 4, 6, 8, 12, 24, 48, 72, 96, 120, 144, and 168 hours postdose on Day 27
Population: All subjects with evaluable concentrations
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Japanese 10 mg | Caucasian 10 mg | Japanese 20 mg | Caucasian 20 mg | Japanese 40 mg | Caucasian 40 mg | Japanese 60 mg | Caucasian 60 mg
Number analyzed (Participants) | 10 | 10 | 6 | 6 | 6 | 6 | 6 | 6
hr | 54.4 (11.0) | 44.3 (7.2) | 40.4 (6.9) | 55.4 (11.5) | 41.6 (8.6) | 39.3 (7.6) | 54.9 (17.4) | 41.8 (9.3)

ADVERSE EVENTS:
Arm/Group | Placebo - Japanese Patients | Placebo - Caucasian Patients | Cohort 1- Japanese Patients | Cohort 1 - Caucasian Patients | Cohort 2 - Japanese Patients | Cohort 2 - Caucasian Patients | Cohort 3 - Japanese Patients | Cohort 3 - Caucasian Patients | Cohort 4 - Japanese Patients | Cohort 4 - Caucasian Patients
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/8 | 0/10 | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/10 | 0/10 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 2/8 | 6/8 | 4/10 | 6/10 | 3/6 | 4/6 | 5/6 | 6/6 | 6/6 | 6/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Japanese Patients (N=8) | Placebo - Caucasian Patients (N=8) | Cohort 1- Japanese Patients (N=10) | Cohort 1 - Caucasian Patients (N=10) | Cohort 2 - Japanese Patients (N=6) | Cohort 2 - Caucasian Patients (N=6) | Cohort 3 - Japanese Patients (N=6) | Cohort 3 - Caucasian Patients (N=6) | Cohort 4 - Japanese Patients (N=6) | Cohort 4 - Caucasian Patients (N=6)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 3 (3) | 5 (5)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Change of Bowel Movement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 4 (4) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mouth Ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 4 (4)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Catheter Site Related Reaction (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thirst (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthropod Bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VIITH Nerve Paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Described in the contract.